CLINICAL TRIAL: NCT04692727
Title: The Effectiveness of Different Taping Methods Applied in Addition to Exercise in Patients With Patellofemoral Pain Syndrome
Brief Title: Taping and Patellar Maltraction in PFPS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ertuğrul Demirdel, Assistant Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/76
Record Dates: First submitted 2020-12-26; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: PFPS; Magnetic Resonance Imaging; McConnell; femoral rotation; taping; malalignment
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Single blind randomized controlled study:Three parallel treatment groups; the control group received only exercise therapy, while the other two groups received two different taping treatments in addition to exercise therapy.
Who Masked: Outcomes Assessor
Masking Description: The information of the individuals being treated will be hidden from the researcher who will make the MRI measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise grup (Active Comparator): An exercise program that includes stretching, strengthening and balance exercises accompanied by physiotherapist in the clinic will be applied to all individuals participating in the study for 6 weeks, 2 times a week (12 sessions). Each session will take approximately 40 minutes and patients will be asked to repeat the exercises at least 2 sets a day at home when they are not in the clinic (other 5 days a week). The home program will be followed by the exercise daily form.
  Interventions: Other: Exercise program
- McConnell patellar taping grup (Experimental): McConnell patellar taping technique will be applied using a rigid tape in addition to the exercise program applied to the exercise group. The tape will remain in the body for a maximum of 48 hours and will be renewed by the same physiotherapist in each session.
  Interventions: Other: Exercise program; Other: McConnel patellar taping technique
- Femoral rotational taping grup (Experimental): Femoral lateral rotation taping technique will be applied using a rigid tape in addition to the exercise program applied to the exercise group.The tape will remain in the body for a maximum of 48 hours and will be renewed by the same physiotherapist in each session.
  Interventions: Other: Exercise program; Other: Femoral rotational taping technique

INTERVENTIONS:
Other: Exercise program — * Hamstring, quadriceps, gastrocnemius, iliopsoas, iliotibial band (ITB), lateral and medial retinaculum stretching exercises
  * Isometric exercises of vastus medialis, gluteus medius and external rotators
  * Isotonic exercises of vastus medialis, gluteus medius and external rotators
  * Closed kinetic chain exercises
  * Balance and coordination exercises
  * Core stabilization exercises
Other: McConnel patellar taping technique — Individuals are placed in a supine position with their knees extended and the quadriceps relaxed. A 5 cm wide hypoallergenic band is applied transversely over the patella without affecting the position of the patella. Then, it is started at the lateral edge of the patella with a rigid tape. The tape is terminated at the medial femoral condyle after a medial pull and / or medial tilt to the patella.
  Arms: McConnell patellar taping grup
Other: Femoral rotational taping technique — This technique is applied in a standing position and hip extreme external rotation. Taping is started on the vastus medialis and is pulled diagonally from the anterior of the leg to the lateral and ends on the trochanter major.
  Arms: Femoral rotational taping grup

SUMMARY:
Patellofemoral Pain Syndrome(PFPS) treatment is basically conservative, but there is no general consensus on the most appropriate therapeutic approach. The aim of this study was to examine the misalignment of the patellofemoral joint with MRI and compare the effectiveness of McConnell patellar taping and femoral lateral rotational taping techniques applied to exercise function on pain, patellar maltraction, functional status, balance and quality of life in patients with PFPS.

DETAILED DESCRIPTION:
This is a single blinded randomized controlled trial, will be conducted at Ankara Yıldırım Beyazıt UniversityYenimahalle Education and Research Hospital. Evaluations regarding the parameters and inclusion criteria at the stage of diagnosis will be carried out by the Specialist Physician, exercise therapy and taping practices by the Specialist Physiotherapist, and the MRI measurements by the Specialist Radiologist. Fixed probability stratified randomization method will be preferred in order to ensure proportional gender distribution in the formation of groups and participants will be divided into 3 groups. An exercise program that includes stretching, strengthening and balance exercises accompanied by physiotherapist in the clinic will be applied to all individuals participating in the study for 2 times/week X 6 weeks (12 sessions). Only the exercise program will be applied to the first group. To the second group; McConnell patellar taping technique will be applied using rigid tape(Leukotape® P Rigid Strapping Tape, 38 mm X 10 m, USA) in addition to the exercise program in each session.To the third group; femoral lateral rotation taping technique will be applied using rigid tape in addition to the exercise program. Patients' patellar maltraction, pain function, balance, and quality of life will be assessed before and after treatment with MRI and clinical testing.

ELIGIBILITY:
Inclusion Criteria:

* Presence of anterior knee pain lasting more than 6 weeks
* Anterior or retropatellar knee pain is present in at least two activities (stair descending, stair climbing, squatting, running, jumping, sitting for a long time
* Presence of malalignment of patellofemoral joint in MRI examination [Bisect offset index (BOİ) ≥57 and / or patellar tilt angle (PTA) ≥15]

Exclusion Criteria:

* presence of knee trauma history and/or previous knee surgery
* presence limitation in knee joint range of motion
* presence of meniscopathy or lesion in knee ligaments
* presence of patellar subluxation or dislocation
* presence of a neuromuscular (upper or lower motor neuron lesions), cardiovascular or rheumatological disease
* pregnancy status
* presence of MRI contraindications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change in Bisect offset index (BOI) | Change from baseline BOI at 6 weeks
  A reference line is drawn through the posterior of the femoral condyles in the axial plan. A line is drawn from the widest diameter of the patella. A perpendicular third line drawn from the deepest point of the trochlear groove divides the widest diameter of the patella into 2 parts (α, β). Bisect offset is defined as the ratio of the lateral part of the patella to the patellar width and is calculated by the formula [α / (α + β) x100]. Being above 57° is a risk factor for pain and patellofemoral joint degeneration.
Change in Patellar tilt angle (PTA) | Change from baseline PTA at 6 weeks
  The patellar tilt angle is the angle between the posterior line of the femoral condyles and the widest mediolateral line of the patella. Below 15 degrees is considered normal.
Change in Lateral patellofemoral angle (LPFA) | Change from baseline LPFA at 6 weeks
  It is the angle between the line connecting the top points of the femoral condyles and the line drawn along the lateral facet of the patella. In general, the patellofemoral angle is more than 8 ° and is open laterally. Medial patency monitoring or an angle less than 8 ° is considered an abnormal slope.
Change in Lateral patellar displacement (LPD) | Change from baseline LPD at 6 weeks
  In the axial plan, a line connecting the top of the medial and lateral condyles and a vertical line is drawn from this at the top of the medial femoral condyle. The distance between this perpendicular line and the medial edge of the patella is measured. This distance should not be more than 1 mm in normal knees.

SECONDARY OUTCOMES:
Visual analog scale (VAS) | Just before the treatment and at the end of 6-week treatment.
  Patients' pain will be assessed for three different situations: "at rest", "at activity" and "at night" before and after treatment. The patient is asked to mark the severity of pain on the 10 cm horizontal line [left end(0) = no pain, right end(10)= unbearable pain ]. Data is measured with a standard ruler and results are recorded in centimeters (cm).
Y balance test (YBT) | Just before the treatment and at the end of 6-week treatment.
  There are 3 bars of 1.5 meters long fixed to a 2.54 cm high central foot plate at an angle of 135 and 90 degrees between them. It is asked to lie down with the tip of the toe in 3 directions and the measurements are recorded.
Kujala Patellofemoral Score (KPS) | Just before the treatment and at the end of 6-week treatment.
  The Kujala Patellofemoral Score developed by Kujala et al contains 13 questions in total. This score questions pain during stair-climbing activity, squatting, running, jumping, and prolonged sitting in knees flexion. It also assesses whether there is disruption, swelling or patellar subluxation, the amount of atrophy in the quadriceps muscle, the presence of flexion deficit, and the need for walking aid. The scoring system ranges from 0 to 100 points, from poor to best . Turkish version of Kujala Patellofemoral Score will be used in individuals with PFPS.
Q angle | Just before the treatment and at the end of 6-week treatment.
  Q angle is the angle formed by a line drawn from the anterosuperior iliac. The angle will be measured in the supine position with the knee in full extension and in two different situations (quadriceps relaxed or maximum voluntary contraction (MVC)).spine to the central patella and a second line drawn from central patella to tibial tubercle.
Nottingham Health Profile (NHP) | Just before the treatment and at the end of 6-week treatment.
  Nottingham Health Profile Questionnaire will be used to evaluate the quality of life. This questionnaire is used to determine how individuals perceive their emotional, social and physical states at that moment. The questions constituting the questionnaire were composed of two options: yes / no. The questionnaire consists of 2 main sections and 6 subtitles (pain, emotional reactions, sleep, social isolation, physical activity, energy) and includes a total of 38 questions. The total score of each section is 100. The scores formed by the answer "Yes" show the negative characteristics of the individual.
Timed up and go test (TUG) | Just before the treatment and at the end of 6-week treatment.
  Patients were asked to perform test at usual walking speed .initial testing standardized verbal instruction given to the participant regarding procedure. For performing TUG participants were instructed to walk three meter and then walk back to sit down .Note time on stopwatch .The average of tests trail was measured as the mean of TUG.
Stair climb test (SCT) | Just before the treatment and at the end of 6-week treatment.
  It is a test that evaluates the patient's staircase up and down activity, lower limb strength, and dynamic balance. The patient is asked to climb up and down 9 steps of 20 cm height as quickly as possible, and the activity time is recorded with a stopwatch. The measurements are repeated 3 times and the average is recorded in seconds.
Genu Valgum/Varum | Just before the treatment and at the end of 6-week treatment.
  The patient is standing. The patient is asked to touch the lower extremities while maintaining knee extension. If the medial condyles are in contact and the distance between the medial malleoli is more than 1 cm, it is evaluated as genu valgum. If the medial malleoli are in contact and the distance between the medial condyles is more than 1 cm, it is considered as genu varum.
Patella type | Just before the treatment and at the end of 6-week treatment.
  Type 1: Medial and lateral facets are concave and almost equal. Type 2: The medial facet is concave and slightly smaller than the lateral facet.
  Type 3: The medial facet is convex and smaller than the lateral facet.
Sulcus angle (SA) | Just before the treatment and at the end of 6-week treatment.
  It is the deepest angle between the medial and lateral trochlear edges. 135 degrees and above are risk factors for patellofemoral osteoarthritis.
Trochlear depth (TD) | Just before the treatment and at the end of 6-week treatment.
  It is measured as the distance from the deepest point of the trochlear sulcus to the line connecting the anterior peaks of the femoral condyles. Below 3 mm is defined as abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Ertuğrul Demirdel, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laugharne E, Bali N, Purushothamdas S, Almallah F, Kundra R. Variability of Measurement of Patellofemoral Indices with Knee Flexion and Quadriceps Contraction: An MRI-Based Anatomical Study. Knee Surg Relat Res. 2016 Dec 1;28(4):297-301. doi: 10.5792/ksrr.16.032. PMID 27894177
- [Background] Nakagawa TH, Muniz TB, Baldon Rde M, Dias Maciel C, de Menezes Reiff RB, Serrao FV. The effect of additional strengthening of hip abductor and lateral rotator muscles in patellofemoral pain syndrome: a randomized controlled pilot study. Clin Rehabil. 2008 Dec;22(12):1051-60. doi: 10.1177/0269215508095357. PMID 19052244
- [Background] Song CY, Huang HY, Chen SC, Lin JJ, Chang AH. Effects of femoral rotational taping on pain, lower extremity kinematics, and muscle activation in female patients with patellofemoral pain. J Sci Med Sport. 2015 Jul;18(4):388-93. doi: 10.1016/j.jsams.2014.07.009. Epub 2014 Jul 24. PMID 25127530
- [Background] Collins NJ, Barton CJ, van Middelkoop M, Callaghan MJ, Rathleff MS, Vicenzino BT, Davis IS, Powers CM, Macri EM, Hart HF, de Oliveira Silva D, Crossley KM. 2018 Consensus statement on exercise therapy and physical interventions (orthoses, taping and manual therapy) to treat patellofemoral pain: recommendations from the 5th International Patellofemoral Pain Research Retreat, Gold Coast, Australia, 2017. Br J Sports Med. 2018 Sep;52(18):1170-1178. doi: 10.1136/bjsports-2018-099397. Epub 2018 Jun 20. PMID 29925502
- [Background] Callaghan MJ, Guney H, Reeves ND, Bailey D, Doslikova K, Maganaris CN, Hodgson R, Felson DT. A knee brace alters patella position in patellofemoral osteoarthritis: a study using weight bearing magnetic resonance imaging. Osteoarthritis Cartilage. 2016 Dec;24(12):2055-2060. doi: 10.1016/j.joca.2016.07.003. Epub 2016 Jul 16. PMID 27432215
- [Background] Callaghan MJ, Selfe J. Patellar taping for patellofemoral pain syndrome in adults. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD006717. doi: 10.1002/14651858.CD006717.pub2. PMID 22513943